CLINICAL TRIAL: NCT01375452
Title: An Open Label, Balanced, Randomized, Two Treatment, Two Sequence, Two Period, Cross-Over, Single-Dose, Comparative Oral Bioavailability Study Of Letrozole 2.5 mg Tablets (Test) of Dr.Reddy's Laboratories Ltd and Femara 2.5 mg Tablets (Reference)of Novartis Pharmaceuticals Corporation, USA In Healthy, Post Menopausal Women Subjects Under Fasting Conditions
Brief Title: Bioavailability Study of Letrozole Tablets 2.5 mg of Dr.Reddy's Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Dr. Ramesh Mullangi -Director, Dr. Reddy's Laboratories Limited
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 032/08
Record Dates: First submitted 2011-06-16; First posted 2011-06-17 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2011-05

CONDITIONS: Healthy
MeSH Terms: interventions — Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Femara (Active Comparator)
  Interventions: Drug: Letrozole
- Letrozole (Experimental)
  Interventions: Drug: Letrozole

INTERVENTIONS:
Drug: Letrozole — Letrozole Tablets 2.5 mg of Dr.Reddy's Laboratories Limited
  Other Names: Femara® Tablets 2.5 mg

SUMMARY:
The purpose of this study is to compare bioavailability in healthy, post menopausal women subjects under fasting conditions.

DETAILED DESCRIPTION:
An Open Label, Balanced, Randomized,Two Treatment, Two Sequence, Two Period, Cross-Over, Single-Dose, Comparative oral bioavailability study in healthy, post menopausal women subjects under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

Healthy post menopausal women within the age range of 40 to 69 years.

* A body mass index within 18-29.9 Kg/m2
* The postmenopausal status should be confirmed by
* Serum Estradiol concentration <40 pg/mL.
* Serum follicle stimulating hormone (FSH) concentration >30 IU/L.
* No vaginal bleeding for at least 1 year.
* Given written informed consent to participate in the study.
* Absence of disease markers of HIV 1 & 2, hepatitis B & C virus and RPR.
* Absence of significant disease or clinically significant abnormal laboratory values on laboratory evaluation, medical history and physical examination during the screening.
* A normal 12-lead ECG.
* A normal chest X-ray (PA view) with in six months before the date of dosing.
* Comprehension of the nature and purpose of the study and compliance with the requirement of the entire protocol.
* No history or no evidence of hypersensitivity/idiosyncratic reaction to Letrozole and related drugs or peanut products or other ingredients of the Letrozole formulation.
* No history of significant systemic diseases.
* Non-smokers.
* No history of psychiatric disorders.
* No donation of blood (one unit or 350 mL) within 56 days prior to study check- in.
* No history of addiction to any recreational drug or drug dependence.
* No participation in any clinical study within the past 56 days.
* No receipt of any prescription drugs within 4 weeks or over-the-counter drugs (e.g.: Cold preparations, and antacid preparations vitamins and natural products used for therapeutic benefits) within 14 days prior to receiving the first dose of study medication or repeated use of drugs within the last four weeks.
* No history of dehydration from diarrhea, vomiting or any other reason within a period of 24 hours prior to study check-in.
* No family history of neurological disorders.
* Not consumed alcohol and xanthine containing food and beverages, (chocolates, tea, coffee or cola drinks) cigarettes and tobacco products, for at least 48 hours, prior to study check-in.
* Not consumed grape fruit containing food or beverages (mosumbi/sweet lime) or poppy containing foods within the 7 days prior to check-in of both the periods.
* Negative results for drugs of abuse (Benzodiazepines, Cocaines, Opioids, Amphetamines, Cannabinoids and Barbiturates) in urine during the each period of study check-in.
* Negative alcohol breathe analysis during the each period of study check-in.

Exclusion Criteria:

The subjects were excluded based on the following criteria.

* Subjects incapable of understanding the informed consent.
* History of suggestive of breast carcinoma, endometrial carcinoma or cervical carcinoma.
* History of suggestive of deep vein thrombosis and/or undiagnosed vaginal bleeding.
* History of thromboembolic disorders.
* History of seizures.
* History of any other major surgical procedure in the past 3 months.
* History of diabetes mellitus and systemic hypertension.
* Past history of anaphylaxis or angioedema.
* History of porphyria, Dubin-Johnson, Rotor syndrome or any other hyperbilirubinemia syndrome.
* History of otosclerosis exacerbated during pregnancy.
* History of cardiovascular, renal, hepatic, ophthalmic, pulmonary, neurological, metabolic,hematological, gastrointestinal, endocrine or immunological diseases.
* Consumption of alcohol for more than two years, or consumption of more than three alcoholic drinks per day or consumption of alcohol within 48 hours prior to dosing and during the study{one drink is equal to one unit of alcohol [one glass wine, half pint beer, and one measure (one ounce) of spirit}.
* History of difficulty with donating blood or difficulty in accessibility of veins.
* An unusual or abnormal diet e.g. low sodium diet, for two weeks prior to receiving any medication and through out subject's participation in the study, for whatever reason e.g. because of fasting due to religious reasons.
* Any major illness in the past three months or any clinically significant ongoing chronic medical illness e.g. congestive heart failure, hepatitis, pancreatitis etc.
* If any Dysplastic changes in the Papanicolaou Smear.
* Female volunteers demonstrating a positive pregnancy test.
* Female volunteers who are currently breast-feeding.
* History of problem in swallowing tablet.
* Used an oral contraceptive containing estrogens or progesterone, or any form of hormonal therapy or intake of HRT and pharmacological agents known to significantly induce or inhibit drug metabolizing enzymes within 6 months of the start of the study.
* History of habituation to coffee, tea or other xanthine containing products and inability to withhold the intake during the-in house-stay.

Ages: 40 Years to 69 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2008-03; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Bioavailability based on Cmax and AUC parameters | 3 Months

CONTACTS AND LOCATIONS:
Overall Officials: A. Jaya Chandra Reddy, FRCS, Principal Investigator — Trident Life Sciences Ltd.